CLINICAL TRIAL: NCT00148187
Title: Prediction of Medication Compliance Following Renal Transplantation
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0202M17442; 2P01DK013083-40A1 (NIH)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Transplantation
Keywords: Medication adherence; Patient compliance; Kidney transplant; Organ rejection; Allograft loss; Drug monitoring
MeSH Terms: conditions — Medication Adherence; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to quantitate pre-transplant medication compliance, dialysis compliance, and related psychological variables, and then examine their validity as predictors of post-transplant noncompliant behaviors and clinically relevant outcomes (acute rejection, graft loss, or death).

Hypothesis: Noncompliance with pre-transplant medication or with the dialysis prescription, and specific psychological variables predict similarly noncompliant behaviors after transplantation.

DETAILED DESCRIPTION:
This pilot study is intended to provide preliminary data about the feasibility of recruiting a cohort of subjects on hemodialysis and following them prospectively through the transplant procedure. The study will document patient adherence to medications and treatment, both before and after surgery. These preliminary data will permit appropriate design and power calculations for a future study assessing our ability to predict post-transplant compliance, based on pre-transplant behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Adult hemodialysis patients in renal transplant evaluation
* Able to read test forms
* Responsible for their own medications

Exclusion Criteria:

* Patients with a major risk of recurrent primary renal disease, e.g. hemolytic uremic syndrome, oxalosis, membranoproliferative glomerulonephritis type II, focal segmental glomerulosclerosis with nephrotic syndrome.
* Patients with active psychosis
* Patients who do not speak English.
* Patients who live and will be followed outside the United States, except Canada.
* Patients who are physically unable to open the Medication Event Monitoring System (MEMS) cap.
* Patients who are not responsible for taking their own medications, e.g. living in a medical care facility.
* Patients who are younger than 14 years old
* Patients who will receive an extra renal organ (except pancreas), either simultaneously or previously.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pre-operative renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2003-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Prediction of early medication adherence | 3 months
  Prediction of declining medication adherence during first three months post kidney transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Nevins, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States